CLINICAL TRIAL: NCT03767959
Title: Evaluation of Chen's U-Suture Technique for Pancreaticojejunostomy Following Pancreaticoduodenectomy
Brief Title: Chen's U-Suture Technique for Pancreaticojejunostomy Following Pancreaticoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C201811
Record Dates: First submitted 2018-11-15; First posted 2018-12-07 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Pancreaticoduodenectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chen's U-Suture (Experimental): Patients in this group will treated by Chen's U-suture technique in pancreaticojejunostomy.
  Interventions: Procedure: Chen's U-Suture
- Classic pancreatic duct to mucosa (Active Comparator): Patients in this group will treated by classic pancreatic duct to mucosa technique in pancreaticojejunostomy.
  Interventions: Procedure: Classic pancreatic duct to mucosa

INTERVENTIONS:
Procedure: Chen's U-Suture — Chen's U-Suture is a new technique of the invaginated end-to-end pancreaticojejunostomy with transpancreatic transverse U-sutures
  Arms: Chen's U-Suture
Procedure: Classic pancreatic duct to mucosa — A Classical anastomosis technique for Pancreaticojejunostomy
  Arms: Classic pancreatic duct to mucosa

SUMMARY:
To date, pancreaticoduodenectomy (PD) is the only recognized potentially curative therapy for malignant neoplasms located in the peri-ampullary region, and is increasingly being used for the treatment of cancer through the resection of the premalignant precursors for invasive carcinomas.Postoperative pancreatic fistula (POPF) is one of the most common complications associated with substantial clinical implications following PD, which significantly affects mortality rate, length of hospital stay, and overall hospital costs. Therefore, the prevention of POPF has always been a high priority for our group as well as other international surgical groups. In 1995, investigators' group established the Chen's U-stitch approach, which was a new technique of end-to-end invaginated pancreaticojejunostomy with transpancreatic transverse U-sutures after PD, and the preliminary results were quite encouraging at that time. Thus, investigators intend to conduct a multicentre, randomized, parallel-group controlled, clinical trial to evaluate the effect and safety of the new technique.

DETAILED DESCRIPTION:
This is a multicentre, randomized, parallel-group controlled, clinical trial to evaluate the effect and safety of Chen's U-Suture technique for pancreaticojejunostomy following pancreaticoduodenectomy. Investigators plan to enroll 960 patients in this study and eligible patients will be randomly divided into two groups. One group will use Chen's U-Suture technique and other group will use classic duct-to-mucosa technique. All patients will be followed up for 3 month after surgery, and primary outcome is POPF, other outcome such as duration of operation, grade of POPF, morbidity, mortality, length of hospital stay, reoperation rate, postoperative pancreatic function and postoperative incidence of chronic pancreatic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 75 years of age, inclusive.
2. Patients have a diagnosis of benign and malignant diseases of the pancreatic head and periampullary region and requiring pancreaticoduodenectomy.
3. Patients have not been treated with any anticancer medications and immunotherapy prior to surgery
4. Patients have not been accompanied by serious physical diseases of heart, lung, brain, etc., and can generally tolerable for surgery.
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Female subjects who are pregnant or breastfeeding.
2. Patients scheduled to undergo pancreatogastrostomy.
3. Patients whose pancreatic duct cannot be located.
4. Patients with history of previous pancreatic surgery, server acute or chronic disease or surgical contraindication.
5. Patients with HIV-infectious or other AIDS-related disease.
6. Patients have any condition that in the judgement of the Investigators would make the subject inappropriate for entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pancreatic Fistula(POPF) | Within 30 days after surgery
  POPF will be strictly classified according to IGSPF criteria

SECONDARY OUTCOMES:
Duration of operation | Intraoperative
  The time of operation count by minute.
Grade of POPF | Within 30 days after surgery
  The grade of POPF will be strictly classified according to IGSPF criteria
Morbidity | Within 90 days after surgery
  The incidence of operative complications within 90 days after surgery.
Mortality | Within 30 days after surgery
  The death occurred within 30 days after surgery
Length of hospital stay after surgery | From first day after surgery to release from hospital (anticipate 5 days minimally)
  Days between surgery and hospital discharge
Reoperation rate | Within one year after surgery
  The incidence of reoperation within 1 year after surgery.
Postoperative pancreatic function | Within one year after surgery
  Postoperative pancreatic function such as blood glucose, blood diastasum diastace, urine amylase, etc.
Postoperative incidence of chronic pancreatic diseases | Within one year after surgery
  The incidence of chronic pancreatic diseases, the chronic pancreatic diseases include chronic pancreatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China